CLINICAL TRIAL: NCT00865280
Title: A Randomized, Evaluator-Blinded, Phase 3 Study to Compare the Safety and Efficacy of PTK 0796 With Linezolid in the Treatment of Adults With Complicated Skin and Skin Structure Infection
Brief Title: Study the Safety and Efficacy of PTK 0796 in Patients With Complicated Skin and Skin Structure Infection (CSSSI)
Acronym: CSSI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated
Sponsor: Paratek Pharmaceuticals Inc (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTK 0796 CSSI-0804
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Results first posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-02

CONDITIONS: Skin Diseases, Infectious
Keywords: CSSI; Abscess; Wound; Cellulitis; Complicated Skin and Skin Structure Infections (cSSSI)
MeSH Terms: conditions — Skin Diseases, Infectious; Abscess; Wounds and Injuries; Cellulitis | interventions — 7-dimethylamino-9-(2,2-dimethylpropyl)aminomethylcycline; omadacycline; Linezolid; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTK 0796 (Experimental): PTK 0796 100 mg for injection; PTK 0796 tablet, 300 mg (2 x 150 mg tablets)
  Interventions: Drug: PTK 0796
- Linezolid (Active Comparator): Gram positive treatment: Linezolid 600 mg tablets and pre-mixed 600 mg IV infusion solution; Gram negative treatment: moxifloxacin 400 mg tablet and moxifloxacin 400 mg IV infusion solution
  Interventions: Drug: linezolid; Drug: moxifloxacin

INTERVENTIONS:
Drug: PTK 0796 — PTK 0796 100 mg for injection; PTK 0796 tablet 150 mg
  Other Names: omadacycline
  Arms: PTK 0796
Drug: linezolid — For gram positive treatment: Linezolid 600 mg tablets and pre-mixed 600 mg IV infusion solution; For gram negative treatment: Moxifloxacin 400 mg tablets and pre-mixed 400mg IV infusion solution
  Other Names: Zyvox™; Avelox™
  Arms: Linezolid
Drug: moxifloxacin — moxifloxacin 400 mg tablet; moxifloxacin 400 mg IV infusion solution
  Arms: Linezolid

SUMMARY:
A Phase III trial to demonstrate the safety and efficacy of PTK 0796 in the treatment of complicated skin and skin structure infections (cSSSI).

DETAILED DESCRIPTION:
The pharmacologic profile of PTK 0796 in humans suggests that it has the potential to be used safely and effectively for this indication. Data from in vitro and animal studies support this hypothesis.

In PTK 0796-CSSI-0804 the safety and efficacy of PTK 0796 in the treatment of cSSSI will be compared to an antibiotic approved for this indication by FDA. Initial treatment will be administered intravenously with the option for subsequent oral treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients, ages 18 years or older
* Is expected to require ≥4 days of IV antibiotic therapy
* Has an acute complicated skin and skin structure infection with findings of systemic inflammatory response
* Female patients must not be pregnant at the time of enrollment and must agree to a reliable method of birth control during the study and for 30 days following the last dose of study drug

Exclusion Criteria:

* Has received an investigational drug within past 1 month
* Has been previously enrolled in this protocol
* Has received >24 hr of a potentially effective systemic antibiotic immediately prior to study drug
* Is nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2009-04-04 (Actual); Primary Completion 2010-04-15 (Actual); Study Completion 2010-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary West, Study Director — Paratek Pharmaceuticals
Locations (7):
- United States (7):
  - Paratek Recruiting Site, Fountain Valley, California
  - Parateck Recruiting Site, La Mesa, California
  - Paratek Recruiting Site, Oceanside, California
  - Paratek Recruiting Site, San Diego, California
  - Paratek Recruiting Site, San Jose, California
  - Parateck Recruiting Site, Columbus, Georgia
  - Paratek Recruiting Site, Savannah, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed to enroll adult participants with Complicated Skin and Skin Structure Infection (CSSI). Participants were stratified at study entry by type of infection (i.e., wound infection, cellulitis, major abscess).
Pre-assignment Details: Participants who met inclusion criteria and did not meet exclusion criteria were randomly assigned to a treatment group.
Groups:
- Omadacycline: Participants received intravenous (IV) omadacycline 100 milligrams (mg) every 24 hours (q24h) for up to 4 to 7 days, then received a 300 mg oral administration q24h. The total treatment duration was up to 14 days. To maintain the blind, participants received an omadacycline infusion alternating with a placebo infusion q12h.
- Linezolid: Participants received IV linezolid 600 mg every 12 hours (q12h) for up to 4 to 7 days, then received a 600 mg oral administration q12h. The total treatment duration was up to 14 days. Participants received moxifloxacin 400 mg q24, IV or oral administration, as appropriate to accompany linezolid for suspected or confirmed gram-negative infections.
Period: Overall Study
Arm/Group | Omadacycline | Linezolid
Started | 70 | 73
Completed | 64 | 70
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 4 | 1
Not completed — End of Treatment/Lost to Follow-up | 0 | 1
Not completed — Adverse Event/Lost to Follow-up | 1 | 0
Not completed — Exclusion Condition | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population: all enrolled participants who received at least one dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Omadacycline | Linezolid | Total
Number analyzed (Participants) | 68 | 72 | 140
Age, Customized [Count of Participants; unit: Participants]
  >=18 to <=44 years | 38 | 51 | 89
  >44 to <=64 | 26 | 20 | 46
  >64 | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 21 | 47
  Male | 42 | 51 | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 56 | 61 | 117
  Black | 7 | 7 | 14
  Asian | 1 | 0 | 1
  Pacific Islander | 2 | 0 | 2
  Other; Not Specified | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified as a Sponsor-defined Clinical Success in the Intent-to-Treat (ITT) Population at End of Treatment
Description: Sponsor-defined clinical success is defined as at least 72 hours of study drug and antibiotics not needed/infection sufficiently resolved. If a participant received antibiotics for a different infection after the primary qualifying infection was considered cured/largely resolved as per the investigator on the Case Report Form (CRF) check box, the participant was also considered as a sponsor-defined clinical success. Sponsor-defined clinical failures must have at least 48 hours of study drug in order to be considered a failure. The sponsor classified participants as clinical failures based on the following: 1) minimum duration of treatment required for outcomes evaluation, 2) use of pre-study antibiotics, 3) use of potentially confounding systemic antibiotics during the study, and 4) timing of concomitant curative surgical procedures.
Time Frame: up to 14 days
Population: Intent-to-Treat (ITT) Population: all enrolled participants who received at least one dose of study medication. Participants were analyzed for efficacy according to randomization, regardless of treatment administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 68 | 72
Participants
  Clinical success | 61 | 66
  Clinical failure | 1 | 3
  Clinical non-evaluable | 6 | 3
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = -2.0, 95% CI 2-sided [-12.4 to 8.5] — The 95% confidence interval (CI) was based on a normal approximation to the binomial distribution with continuity correction. Treatment difference for a response of clinical success was calculated as omadacycline minus linezolid

2. Primary Outcome: Number of Participants Classified as a Sponsor-defined Clinical Success in the ITT Population at Test of Cure
Description: Sponsor-defined clinical success is defined as at least 72 hours of study drug and antibiotics not needed/infection sufficiently resolved. If a participant received antibiotics for a different infection after the primary qualifying infection was considered cured/largely resolved as per the investigator on the CRF check box, the participant was also considered as a sponsor-defined clinical success. Sponsor-defined clinical failures must have at least 48 hours of study drug in order to be considered a failure. The sponsor classified participants as clinical failures based on the following: 1) minimum duration of treatment required for outcomes evaluation, 2) use of pre-study antibiotics, 3) use of potentially confounding systemic antibiotics during the study, and 4) timing of concomitant curative surgical procedures.
Time Frame: 10 to 17 days after last dose of treatment (total treatment of up to 14 days)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 68 | 72
Participants
  Clinical success | 58 | 64
  Clinical failure | 2 | 3
  Clinical non-evaluable | 8 | 5
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = -3.6, 95% CI 2-sided [-15.5 to 8.3] — The 95% CI was based on a normal approximation to the binomial distribution with continuity correction. Treatment difference for a response of clinical success was calculated as omadacycline minus linezolid

3. Primary Outcome: Number of Participants With Wound Infections Classified as a Sponsor-defined Clinical Success in the Clinically Evaluable (CE) Population at End of Treatment
Description: as for outcome 2
Time Frame: up to 14 days
Population: CE Population: all participants in the ITT Population who met specific criteria such that the clinical outcome of their infection could be inferred to reflect the effect of the study drug. Only those participants stratified with wound infection at study entry were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 13 | 13
Participants
  Clinical success | 13 | 12
  Cinical failure | 0 | 1
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = 7.7, 95% CI 2-sided [-11.2 to 26.6] — [estimate comment as in outcome 2, analysis 1]

4. Primary Outcome: Number of Participants With Cellulitis Classified as a Sponsor-defined Clinical Success in the CE Population at End of Treatment
Description: as for outcome 2
Time Frame: up to 14 days
Population: CE Population: all participants in the ITT Population who met specific criteria such that the clinical outcome of their infection could be inferred to reflect the effect of the study drug. Only those participants stratified with cellulitis at study entry were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 39 | 45
Participants
  Clinical success | 38 | 44
  Clinical failure | 1 | 1
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = -0.3, 95% CI 2-sided [-8.3 to 7.6] — [estimate comment as in outcome 2, analysis 1]

5. Primary Outcome: Number of Participants With Wound Infections Classified as a Sponsor-defined Clinical Success in the CE Population at Test of Cure
Description: as for outcome 2
Time Frame: 10 to 17 days after last dose of treatment (total treatment of up to 14 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 13 | 13
Participants
  Clinical success | 13 | 12
  Clinical failure | 0 | 1
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = 7.7, 95% CI 2-sided [-11.2 to 26.6] — [estimate comment as in outcome 2, analysis 1]

6. Primary Outcome: Number of Participants With Cellulitis Classified as a Sponsor-defined Clinical Success in the CE Population at Test of Cure
Description: as for outcome 2
Time Frame: 10 to 17 days after last dose of treatment (total treatment of up to 14 days)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 39 | 45
Participants
  Clinical success | 38 | 44
  Clinical failure | 1 | 1
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = -0.3, 95% CI 2-sided [-8.3 to 7.6] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Number of Participants With the Indicated Type of Adverse Event (AE)
Description: The assessment of safety was based mainly on the frequency of AEs, and summaries of vital signs and laboratory values (values classified as AE are captured in the AE module). An AE is defined as the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug, whether or not the event was considered causally related to the medical product. An AE could have been a new occurrence or an existing process that increased in intensity or frequency. AEs were deemed treatment-emergent if the start date was on or after the date of the first dose but was not present before that date or if the AE started before the date of the first dose and increased in severity on or after that date.
Time Frame: from the time of informed consent to Test of Cure (10 to 17 days after end of treatment [total treatment of up to 14 days)
Population: Safety Population: all enrolled participants who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 68 | 72
Participants
  Treatment-emergent adverse event (TEAE) | 56 | 58
  Study drug-related TEAE | 41 | 41
  AEs leading to study drug discontinuation | 2 | 0

ADVERSE EVENTS:
Time Frame: from the time of informed consent to Test of Cure (10 to 17 days after end of treatment [total treatment of up to 14 days])
Description: Adverse events are reported for members of the Safety Population, comprised of all enrolled participants who received at least one dose of study medication
Arm/Group | Omadacycline | Linezolid
All-Cause Mortality (participants affected / at risk) | 1/68 | 0/72
Serious Adverse Events (participants affected / at risk) | 3/68 | 1/72
Other Adverse Events (participants affected / at risk) | 52/68 | 55/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline (N=68) | Linezolid (N=72)
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline (N=68) | Linezolid (N=72)
Palpitations (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 18 | 19
Constipation (Gastrointestinal disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 6 | 11
Diarrhoea (Gastrointestinal disorders) | 3 | 13
Dry mouth (Gastrointestinal disorders) | 3 | 1
Toothache (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Infusion site pain (General disorders) | 5 | 2
Fatigue (General disorders) | 3 | 3
Infusion site erythema (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 3 | 1
Cellulitis (Infections and infestations) | 2 | 1
Infection (Infections and infestations) | 2 | 1
Abscess (Infections and infestations) | 1 | 2
Oral candidiasis (Infections and infestations) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 6 | 2
Alanine aminotransferase increased (Investigations) | 1 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 2
Increased appetite (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 16 | 5
Dizziness (Nervous system disorders) | 7 | 6
Dysgeusia (Nervous system disorders) | 1 | 4
Insomnia (Psychiatric disorders) | 2 | 5
Dysuria (Renal and urinary disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 6
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2
Flushing (Vascular disorders) | 2 | 0
Pain (General disorders) | 2 | 1
Tremor (Nervous system disorders) | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
Changes in Food and Drug Administration (FDA) criteria for the identification and enrollment of participants with complicated skin and skin structure infections as well as the primary endpoint led to administrative termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less